CLINICAL TRIAL: NCT06148311
Title: Dexmedetomidine Sublingual Film for the Ambulatory Treatment of Hyperadrenergic Autonomic Crisis in Patients With Familial Dysautonomia
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-01332; 1R01FD007826-01 (FDA)
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Familial Dysautonomia
Keywords: Familial Dysautonomia; Hereditary Sensory and Autonomic Neuropathy type 3; HSAN; autonomic sympathetic crises
MeSH Terms: conditions — Dysautonomia, Familial; Hereditary Sensory and Autonomic Neuropathies | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sublingual dexmedetomidine (Experimental): Participants will be administered 120 micrograms sublingual film following start of an autonomic crisis. In case the crisis has not subsided after 2 hours, the patient will be instructed to take the second dose. The maximum amount for the study is two oral films within two hours for each episode but not more than 24 hours apart, one at the beginning of the crisis and if needed, one additional within two hours.
  Interventions: Drug: Dexmedetomidine
- Matching Sublingual Placebo (Placebo Comparator): Participants will be administered the matching placebo sublingual film following start of an autonomic crisis. In case the crisis has not subsided after 2 hours, the patient will be instructed to take the second dose. The maximum amount for the study is two oral films within two hours for each episode but not more than 24 hours apart, one at the beginning of the crisis and if needed, one additional within two hours.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Matching placebo — One matching placebo will be given under the tongue on a thin dissolvable film.
  Arms: Matching Sublingual Placebo
Drug: Dexmedetomidine — Dexmedetomidine 120 mcg will be given under the tongue on a thin dissolvable film.
  Arms: Sublingual dexmedetomidine

SUMMARY:
The purpose of this placebo controlled interventional study is to collect preliminary data on administering dexmedetomidine in patients with Familial Dysautonomia (FD) during a rapid cessation of autonomic crisis. The primary aims are to assess the feasibility and evaluate if measurements of heart rate, blood pressure and oxygen saturation can predict the start of an autonomic crisis.

Funding Source- FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of Familial Dysautonomia.
* One or more autonomic crises during the last year.
* Our database shows evidence of autonomic crisis, previous treatment with IV dexmedetomidine, and registered medical data within the year preceding the study.
* Age 16 years or older
* The patient has a responsible caretaker to communicate with the medical providers.
* Provision of signed and dated informed consent form from the patient and responsible caregiver
* Able to state willingness to comply with all study procedures and availability for the duration of the study
* For males and females of reproductive age: use condoms for contraception if sexually active.

Exclusion Criteria:

* At the consideration of the principal investigator, the caregiver cannot fully understand the protocol, or communicate during the crisis with the Center.
* The patient during the crisis, before taking the medication, has any of the following:

  1. Oxygen saturation less than 92% on room air or baseline need for oxygen, change from baseline oxygen dependency.
  2. Respiratory rate >25 breaths per minute.
  3. Supine blood pressure ≤ 90/860mmHg
  4. Febrile illness with temperature >100.3 F.
  5. Serological signs of infection (WBC count >10 g/dL, or CRP >10 mg/L or ESR>20, or above their steady historical baseline levels) in recent (less than one month) studies.
* The patient is a female and has a positive pregnancy test.
* The Montreal Cognitive Exam (MoCA) is below 25 points.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with reduction of Autonomic crisis severity assessment scores (ACSAS) to ≤ 5 points | Up to 2 hours post administration
  ACSAS tool will be used to measure objectively and record signs and symptoms of autonomic crisis, which includes documentation of blood pressure, heart rate, skin flushing and blotching, sweating, and behavioral changes. Scores are totaled at each timepoint (0 minutes, 15 min., 45 min., 1.5 hours, 2hr.) ranging from 0 (Normal) to 16 (most severe symptoms occurred).
Percentage of patients with 25% reduction in blood pressure | Up to 2 hours post administration
  Patients will be monitored with a hospital-at-home (H@H) device to allow visualization of vital signs in real life. The H@H monitor (Biobeat™) is an FDA approved device and will be attached to the patient´s chest by an adhesive patch which will transmit blood pressure. Blood pressure will be monitored before taking each dose and up to 2 hours after.
Percentage of patients with >20% reduction in heart rate | Up to 2 hours post administration
  Patients will be monitored with a hospital-at-home (H@H) device to allow visualization of vital signs in real life. The H@H monitor (Biobeat™) is an FDA approved device and will be attached to the patient´s chest by an adhesive patch which will transmit heart rate. Heart rate will be monitored before taking each dose and up to 2 hours after.
Percentage of patients with >50% reduction in vomiting/retching episodes | Up to 2 hours post administration
  Patients will be monitored by their care givers for of episodes of vomiting/ retching before taking each dose and up to 2 hours after.

SECONDARY OUTCOMES:
Percentage of patients with ≥ 20% reduction in hospitalizations | Up to 48 months
  Study team will compare historical data to number of hospitalizations occurred after taking one or more doses.
Percentage of patients with ≥ 20% reduction in hospital stay duration | Up to 48 months
  Study team will compare historical data to number of days during hospital stay that occurred after taking one or more doses.
Percentage of patients with ≥ 30% reduction in ICU stay duration | Up to 48 months
  Study team will compare historical data to number of days at the ICU that occurred after taking one or more doses.
Change in number of medical complications | Baseline, up to 48 months
  Study team will compare historical data to number of medical complications of hospitalizations occurred after taking one or more doses.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Gonzalez-Duarte, MD, Principal Investigator — NYU Langone Health, NYU Dysautonomia Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Alejandra.gonzalez-duarte@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Alejandra.gonzalez-duarte@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.